CLINICAL TRIAL: NCT03614897
Title: Prevention of Falls in the Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1712-62
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Accidental Falls
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Experimental): Providers participating in education related to guidelines for treating patients at risk of falling
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Education on guidelines for care of individuals at risk of falling

SUMMARY:
An educational intervention will be utilized to improve care following guidelines for treating individuals at risk of falling. A survey will be administered to providers pre and post education.

ELIGIBILITY:
Inclusion Criteria:

* Primary care providers in Family Medicine and Internal Medicine

Exclusion Criteria:

* Providers in outlying clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Harbison, DO, Principal Investigator — The Guthrie Clinic; Sheela Prabhu, MD, Principal Investigator — The Guthrie Clinic
Locations (1):
- Guthrie Medical Group, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harbison AJ, Prabhu S. Causation and Treatment Algorithms for Elderly Patients who have Fallen in the Twin Tiers. Cureus. 2019 Dec 30;11(12):e6513. doi: 10.7759/cureus.6513. PMID 32025432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical providers in internal medicine and family medicine were surveyed
Groups:
- Education: Providers were offered an educational program focusing on the guidelines. A survey was completed prior to the presentation and one year after.
Period: Overall Study
Arm/Group | Education
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Education
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender is unknown due to anonymous survey
  Participants
    Unknown | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Survey Score for Providers' Self-reported View on Vitamin Deficiency as a Cause of Falls
Description: Absolute change in mean survey score before and after education for providers' view on vitamin D deficiency as a cause of falls. The scale is a likert scale from 1-5: 1 important, 2 somewhat important, 3 neither important nor important, 4 somewhat important, 5 unimportant.
Time Frame: 1year
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-education: Provider survey responses before education
- Post-education: Provider survey responses after education
Arm/Group | Pre-education | Post-education
Number analyzed (Participants) | 43 | 42
score on a scale | 4.23 (0.51) | 3.44 (0.96)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Groups:
- Education: Providers were offered an educational program focusing on the guidelines.
  A survey was completed prior to the presentation and one year after.
  The medical records for 1 year post education were reviewed for falls and compliance to the guidelines.
Arm/Group | Education
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03614897/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT03614897/SAP_001.pdf